CLINICAL TRIAL: NCT06826482
Title: Evaluation of the Effects of Tongue-Tie and Upper Lip-Tie on Breastfeeding With Ultrasound Measurements and the LATCH Breastfeeding Assessment Tool
Brief Title: Evaluation of the Effects of Tongue-Tie and Upper Lip-Tie
Status: Completed | Type: Observational
Sponsor: Ankara Yildirim Beyazıt University (Other)
Responsible Party: Sponsor
Other Study IDs: 26379996/06
Record Dates: First submitted 2025-02-01; First posted 2025-02-14 (Actual); Last update posted 2025-02-14 (Actual); Status verified 2025-02

CONDITIONS: Tongue-tie; Upper Lip-tie
Keywords: Tongue-tie; upper lip-tie; breastfeeding; ultrasonography; newborn
MeSH Terms: conditions — Ankyloglossia; lip tie; Breast Feeding

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- tongue-tie: To evaluate the tongue and lingual frenulum, the TABBY assessment tool, which consists of 12 images demonstrating the appearance of the tongue tip, the insertion of the frenulum, and the mobility of the tongue (lift and protrusion), was used. It has a score between 0 and 8. Normal tongue function is represented by a score of 8; borderline values are represented by scores of 6 and 7; and impaired tongue function is indicated by scores of 5 and below. Newborns who scored five or below were included in the tongue-tie group.
- upper lip-tie: The maxillary labial frenulum in the newborn was examined by lifting the upper lip and classified according to Kotlow. Newborns with a frenulum grade 3 (the frenulum inserts just in front of the anterior papilla) or grade 4 (the frenulum attaches just into the anterior papilla and extends into the hard palate) were included in the upper lip-tie group.
- control: The control group comprised newborns without tongue-tie or upper lip-tie

SUMMARY:
Background: Tongue-tie and upper-lip tie have been linked to breastfeeding difficulties; however, the traditional evaluation tools that provide this information rely primarily on subjective assessments. In this context, ultrasound imaging has enabled an objective assessment of the sucking dynamics of infants. The aim of this study was to assess the impact of tongue-tie and upper lip-tie on sucking function in newborns via ultrasonography and other tools.

Methods: This prospective cohort study included 67 newborns (25 with tongue-tie, 21 with upper lip-tie, and 21 control) as well as their mothers. The maxillary labial frenulum was evaluated according to Kotlow, and the lingual frenulum was evaluated according to the Tongue Tie and Breastfed Infants (TABBY) tool. Sucking functions were examined via ultrasonography between postnatal days 5 and 15. Breastfeeding was evaluated via the LATCH tool, and maternal nipple pain was graded via a numerical rating scale. Mothers were interviewed by telephone about their breastfeeding continuity in the 1st month after birth. The data were analyzed through descriptive and inferential statistics and association tests.

DETAILED DESCRIPTION:
1. Sample characteristics and study design:

   This prospective cohort study was conducted at Ankara Yıldırım Beyazit University Faculty of Medicine, Internal Medicine Sciences, Department of Child Health and Diseases, Neonatology Clinic, from May 2022 to December 2022. The study included newborns with tongue-tie, newborns with upper lip-tie, and newborns without both. Written informed consent was obtained from all participating mothers, and the study was approved by the Clinical Research Ethics Committee of Ankara Yıldırım Beyazit University Faculty of Medicine (date and number: 30.03.2022 /26379996/06).

   The inclusion criteria were breastfed newborns born within the last 48 hours, with a gestational age of 38 weeks or more, uncomplicated delivery, and no systemic problems, craniofacial anomalies, or birth defects. The exclusion criteria included premature or low birth weight newborns; those with delivery complications; intensive care unit admissions; systemic problems; craniofacial anomalies; birth defects; both tongue-tie and upper lip-tie; and those exclusively formula-fed.

   As there was no comparable study that could be consulted to determine the sample size in the literature, a total of 60 neonates were recruited, with 20 in each group: tongue-tie (group 1), upper lip-tie (group 2), and control (group 3).
2. Data collection:

   Data on maternal age, medical conditions, pregnancy medication, consanguineous marriage, number of births, breastfeeding experience, and breastfeeding education were collected via face-to-face interviews. Gestational week, sex, birth weight and mode of delivery were obtained from the birth records.

   The baby's tongue movements while crying were observed for lingual frenulum examination. To evaluate the tongue and lingual frenulum, the TABBY assessment tool, which consists of 12 images demonstrating the appearance of the tongue tip, the insertion of the frenulum, and the mobility of the tongue (lift and protrusion), was used. It has a score between 0 and 8. Normal tongue function is represented by a score of 8; borderline values are represented by scores of 6 and 7; and impaired tongue function is indicated by scores of 5 and below. Newborns who scored five or below were included in the tongue-tie group in this study.

   The maxillary labial frenulum in the newborn was examined by lifting the upper lip and classified according to Kotlow [4]. Newborns with a frenulum grade 3 (the frenulum inserts just in front of the anterior papilla) or grade 4 (the frenulum attaches just into the anterior papilla and extends into the hard palate) were included in the upper lip-tie group. In addition, when the upper lip was lifted upward, whether the upper lip touched the newborn's nose and whether whitening occurred in the area where the frenulum adhered to the alveolar crest were noted.

   The control group comprised newborns without tongue-tie or upper lip-tie.

   Ultrasound imaging was conducted between the 5th and 15th days after birth by a single dentomaxillofacial radiologist with 14 years of experience. To evaluate the infants' sucking abilities, the mother was seated in a comfortable chair in the correct posture for breastfeeding. A GE Medical System Verasana Active (Wuxi, Jiangsu, China) mobile ultrasonography device equipped with a 6-10 MHz 8C-RS microconvex probe was used to capture 2D real-time, B-mode, and M-mode images of the oral cavity of the neonates. Imaging was performed through a submental approach via ultrasonic gel (Aquasonic, Parker Labs., Fairfield, NJ, USA).

   The data collection commenced when the infant began to latch onto the breast and concluded when the feeding ended. The study excluded recordings that exhibited artifacts resulting from movements of the mother-newborn pair or the operator, as well as recordings in which the presence of nutritive sucking could not be observed. All measurements were conducted on recorded ultrasonography images. Before starting the measurement in the study, the observer was calibrated to recognize and identify the neonate maxillofacial and oral anatomy; for this purpose, 10 different neonate ultrasonography images other than those used in the study were used. The observer was blinded to any patient data.

   During sucking, ultrasound imaging of the tongue, hyoid bone, nipple, and hard and soft palates was performed in the midsagittal plane. A suck cycle was defined as beginning when the mid-tongue was in apposition with the palate (tongue up), followed by a downward excursion of the tongue until the mid-tongue reached its lowest point (tongue down) and then reunited with the palate. During sucking, while the tongue is positioned both upward and downward, the distance between the nipple (N) and the hard-soft palate junction (HSPJ), the depth of the intraoral space (the distance from the HSPJ to the surface of the mid-tongue), the nipple diameter (ND) measured at intervals of 2, 5, 10, and 15 mm from the tip of the nipple, and the anterior and mid-tongue heights (the distance between the dorsal surface of the anterior and mid-tongues and the inferior border of the genioglossus muscle) were assessed via ultrasound imaging.

   Breastfeeding was assessed via the LATCH tool during ultrasound imaging. This tool consists of 5 items that score latch, audible swallowing, type of nipple, comfort, and hold (positioning). Each item is evaluated on a scale of 0-2 points. The highest possible total score that can be obtained from the LATCH assessment tool is 10. A high score indicates greater success in breastfeeding.

   To evaluate nipple pain, the mother was asked to rate her pain during breastfeeding on a numerical scale. A score of 0 indicated "absence of pain," and a score of 10 indicated "presence of unbearable pain".

   Newborns' feeding practices (exclusive or nonexclusive breastfeeding) were also noted.

   Mothers were interviewed by telephone at the 1st month after birth and asked questions about infant feeding practices, maternal nipple pain, and whether any intervention was made for newborns with tongue-tie and upper lip-tie.
3. Statistical analysis:

The data were analyzed via IBM SPSS Statistics 22.0 (IBM SPSS Statistics for Windows, Version 22.0. Armonk, NY: IBM Corp) Nonnormally distributed data were compared via the Mann-Whitney U test for paired groups and the Kruskall-Wallis H test for three or more groups. Descriptive statistics, chi-square test and correlation analyses were conducted. A value of p<0.05 was considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* Breastfed newborns born within the last 48 hours
* Gestational age of 38 weeks or more
* Uncomplicated delivery
* Absence of systemic problems, craniofacial anomalies, or birth defects.

Exclusion Criteria:

* Premature or low birth weight newborns
* Newborns with delivery complications
* Newborns admitted to the intensive care unit
* Any systemic problems, craniofacial anomalies, birth defects
* Presence of both tongue-tie and upper lip-tie
* Newborns exclusively formula-fed.

Ages: 1 Hour to 48 Hours | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Newborns born within the last 48 hours
Sampling Method: Non-Probability Sample
Enrollment: 67 (Actual)
Dates: Start 2022-05-01 (Actual); Primary Completion 2022-12-01 (Actual); Study Completion 2022-12-01 (Actual)

PRIMARY OUTCOMES:
Distance between the nipple (N) and the hard-soft palate junction | Between the 5th and 15th days after birth.
  During sucking, while the tongue is positioned both upward and downward, the distance between the nipple (N) and the hard-soft palate junction (HSPJ) was measured via ultrasound imaging.
Intraoral space dept | Between the 5th and 15th days after birth.
  During sucking, while the tongue is positioned both upward and downward, the intraoral space dept (the distance from the HSPJ to the surface of the mid-tongue) was measured via ultrasound imaging.
Nipple diameter (ND) at 2 mm from the tip of the nipple. | Between the 5th and 15th days after birth.
  During sucking, while the tongue is positioned both upward and downward, the nipple diameter (ND) at 2 mm from the tip of the nipple was measured via ultrasound imaging.
Nipple diameter (ND) at 5 mm from the tip of the nipple. | Between the 5th and 15th days after birth.
  During sucking, while the tongue is positioned both upward and downward, the nipple diameter (ND) at 5 mm from the tip of the nipple was measured via ultrasound imaging.
Nipple diameter (ND) at 10 mm from the tip of the nipple. | Between the 5th and 15th days after birth.
  During sucking, while the tongue is positioned both upward and downward, the nipple diameter (ND) at 10 mm from the tip of the nipple was measured via ultrasound imaging.
Nipple diameter (ND) at 15 mm from the tip of the nipple. | Between the 5th and 15th days after birth.
  During sucking, while the tongue is positioned both upward and downward, the nipple diameter (ND) at 15 mm from the tip of the nipple was measured via ultrasound imaging.
Anterior-tongue height | Between the 5th and 15th days after birth.
  During sucking, while the tongue is positioned both upward and downward, the anterior-tongue height (the distance between the dorsal surface of the anterior-tongue and the inferior border of the genioglossus muscle) was measured via ultrasound imaging.
Mid-tongue height | Between the 5th and 15th days after birth.
  During sucking, while the tongue is positioned both upward and downward, the mid-tongue height (the distance between the dorsal surface of the mid-tongue and the inferior border of the genioglossus muscle) was measured via ultrasound imaging.
LATCH scores | Between the 5th and 15th days after birth (at the ultrasound appointment)
  Breastfeeding was assessed via the LATCH tool. This tool consists of 5 items that score latch, audible swallowing, type of nipple, comfort, and hold (positioning). Each item is evaluated on a scale of 0-2 points. The highest possible total score that can be obtained from the LATCH assessment tool is 10. A high score indicates greater success in breastfeeding.
Maternal nipple pain | Between the 5th and 15th days after birth (at the ultrasound appointment) and the 1st month after birth (questioned at a telephone interview).
  Maternal nipple pain was graded via a numerical rating scale. A score of 0 indicated "absence of pain," and a score of 10 indicated "presence of unbearable pain".

OTHER OUTCOMES:
Maternal age | Baseline
  Maternal age was recorded.
Maternal chronic diseases | Baseline
  The medical condition of the mother was recorded.
Maternal medication use | Baseline
  Presence or absence of medication during pregnancy was recorded.
Consanguineous marriage | Baseline
  Presence or absence of consanguineous marriage was recorded.
Number of births by mother | Baseline
  The number of births by the mother was recorded.
Breastfeeding experience | Baseline
  Presence or absence of breastfeeding experience was recorded.
Breastfeeding education | Baseline
  Presence or absence of breastfeeding education was recorded.
Gestational week | Baseline
  Gestational week was obtained from the birth records.
Gender | Baseline
  The Gender of the newborn was obtained from the birth records.
Birth weight | Baseline
  The birth weight (in grams) of the newborn was obtained from the birth records.
Mode of delivery | Baseline
  The mode of delivery (vaginal or cesarean) was obtained from the birth records.
Newborns' feeding practices | Between the 5th and 15th days after birth (at the ultrasound appointment) and the 1st month after birth (questioned at a telephone interview).
  Newborns' feeding practices were recorded as exclusive or nonexclusive breastfeeding.
Surgical Intervention (Frenotomy) | 1st month after birth (questioned at a telephone interview).
  Presence or absence of surgical intervention for the frenulum was recorded.

CONTACTS AND LOCATIONS:
Locations (2):
- Turkey (Türkiye) (2):
  - Ayse Isil Orhan, Ankara
  - Department of Pediatric Dentistry, Faculty of Dentistry, Ankara Yildirim Beyazit University,, Ankara

IPD SHARING:
Plan to Share IPD: No